CLINICAL TRIAL: NCT04710771
Title: Effect of Prone Positioning and Alternate Nostril Breathing Technique in Patients With COVID-19: A Quasi Experimental Study.
Brief Title: Effect of Prone Positioning in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sialkott College of Physical Therapy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 138-2020
Record Dates: First submitted 2021-01-09; First posted 2021-01-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Covid19
Keywords: Covid-19; General Anxiety Disorder-7; Prone Position; Alternate Nostril Breathing
MeSH Terms: conditions — COVID-19 | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Experimental): Patient performed prone lying position for three hours.
  Interventions: Other: Prone Lying Position
- Group-B (Active Comparator): along with Prone lying position, patients also performed alternate nostril breathing for ten minutes.
  Interventions: Other: Prone Lying Position; Other: alternate nostril breathing

INTERVENTIONS:
Other: Prone Lying Position — patient lies on his/ her stomach facing floor.
  Other Names: Positioning
Other: alternate nostril breathing — patient inspires with one nostril at a time, right or left one by one and expires by mouth.
  Other Names: breathing technique
  Arms: Group-B

SUMMARY:
COVID-19 is affecting the people around the world and the infected individuals' may either stay asymptomatic or present to hospitals with severe distress and life threatening symptoms. The objective of the study is to investigate role of Prone positioning and alternate nostril breathing in patients with Covid-19.

DETAILED DESCRIPTION:
In this quasi experimental study, 30 patients aged 40-80 years of either gender with a confirmed diagnosis of COVID-19 receiving supplemental oxygen were recruited from DHQ Hospital Faisalabad. patients were grouped into two A & B. We collected baseline data on demographics and anthropometrics. After baseline data collection, all the patients were helped into the prone position, which was maintained for a minimum duration of three hours. After that patients in group B performed alternate nostril breathing for 10 minutes with help of physiotherapist. Clinical data were re-collected on 3rd day of intervention one hour after returning to the supine position in group A and after alternate nostril breathing in group B. The main study outcome was the variation in oxygenation (partial pressure of oxygen [PaO2]/ fractional concentration of oxygen in inspired air [FiO2]) between baseline and resupination, and General psychological state through GAD-7 General anxiety disorder questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Age: 40-80 Gender: Both GCS score:15

Exclusion Criteria:

* COPD Intubated ARDS Smoker Neurological Disorder

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
PaO2 | Change in score before the intervention on 1st day of intervention and on 3rd day one hour after the intervention.
  partial pressure of oxygen.
FiO2 | Change in score before the intervention on 1st day of intervention and on 3rd day one hour after the intervention.
  Fractional concentration of oxygen in inspired air [FiO2])
General Anxiety Disorder-7 Score | Change in score before the intervention on 1st day of intervention and on 3rd day one hour after the intervention.
  general anxiety disorder-7 score ranges from 0-21, out of which 0-4 means minimal anxiety, 5-9 stands for mild anxiety, 10-14 for moderate and 15-21 for severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sahreen Anwar, PhD, Principal Investigator — Independent Medical College, Faisalabad
Locations (1):
- DHQ Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No